CLINICAL TRIAL: NCT00647478
Title: A Multicenter Study to Assess Differences Between Circulating Levels of IGF-I and IGFBP-3 in Patients With Sporadic Late-onset Alzheimer's Disease and Control Elderly Subjects.
Brief Title: System-IGF-1 Pathway and Alzheimer's Disease
Acronym: SIGAL
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: P060224
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment; Cognitive Function 1, Social; Control With Normal Activities of Daily Living
Keywords: Insulin-like Growth Factor; Insulin-like Growth Factor binding protein 3; Insulin-like Growth Factor-I system component levels; Insulin-like Growth Factor-I polymorphism; Alzheimer's disease; Mild Cognitive Impairment; Normal cognitive function; Observational cross sectional study
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for plasma levels and polymorphisms in IGF1 system components
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: AD
- 2: Control elderly subjects with normal cognitive function
- 3: MCI

SUMMARY:
The aim is to assess the relationship between levels of IGF-I system components and cognitive status in patients with Alzheimer's disease (AD), in elderly subjects with normal cognitive function, and in patients with mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
AD is the most common cause of dementia. During aging, decline of biological brain functions due to a number of genetic and environmental factors facilitates the onset of AD. MCI includes prodromal AD.

The identification of the risk factors for AD must be a priority in order to define the best therapeutic approach.

Recent data support the notion that IGF-I pathway accounts for neuronal protection, with a dual effect, on both brain Aβ peptide and tau protein.

This large, multicenter, prospective, observational, cross-sectional population-based study in 3 parallel groups (200 participants per group) is aimed to assess differences between IGF-I and IGFBP3 circulating levels and polymorphisms in AD patients and control elderly subjects, and in MCI patients.

ELIGIBILITY:
Inclusion Criteria:

Caucasian patients after a comprehensive geriatric assessment and giving informed written consent.

- In each arm :

1. elderly subjects with normal cognitive function,
2. patients with dementia of AD type (DSM-IV and NINCDS-ADRDA criteria),
3. patients with MCI (European Consortium on Alzheimer's Disease, EADC).

Exclusion Criteria:

Non AD dementia Major depression Use of anticholinesterase agent All diseases or major sensory deficits or any condition that might interfere with cognitive assessment and study objectives

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Ambulatory Elderly subjects
Sampling Method: Non-Probability Sample
Enrollment: 693 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Circulating IGF-I and IGFBP-3 levels in AD patients and control elderly subjects at the time of assessment(T0). | 24 hours

SECONDARY OUTCOMES:
Circulating IGF-I and IGFBP-3 levels | 24 hours
Genetic polymorphisms in IGF-I / IGFBP-3 | 24 hours
Circulating IGF-I and IGFBP-3 levels and genetic polymorphisms in IGF-I / IGFBP-3 according to cognitive function. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hanon, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Broca Hospital Memory Clinic (CMRR), Paris, Paris, France

REFERENCES:
- [Background] Murialdo G, Barreca A, Nobili F, Rollero A, Timossi G, Gianelli MV, Copello F, Rodriguez G, Polleri A. Relationships between cortisol, dehydroepiandrosterone sulphate and insulin-like growth factor-I system in dementia. J Endocrinol Invest. 2001 Mar;24(3):139-46. doi: 10.1007/BF03343833. PMID 11314741
- [Background] Duron E, Vidal JS, Funalot B, Brunel N, Viollet C, Rigaud AS, Labouree F, Epelbaum J, le Bouc Y, Hanon O. Insulin-Like Growth Factor-I, Insulin-Like Growth factor Binding Protein-3 and Blood Hemoglobin Concentration in an Elderly Population. J Gerontol A Biol Sci Med Sci. 2015 Jul;70(7):854-9. doi: 10.1093/gerona/glu200. Epub 2014 Nov 9. PMID 25384548
- [Background] Duron E, Funalot B, Brunel N, Coste J, Quinquis L, Viollet C, Belmin J, Jouanny P, Pasquier F, Treluyer JM, Epelbaum J, le Bouc Y, Hanon O. Insulin-like growth factor-I and insulin-like growth factor binding protein-3 in Alzheimer's disease. J Clin Endocrinol Metab. 2012 Dec;97(12):4673-81. doi: 10.1210/jc.2012-2063. Epub 2012 Sep 26. PMID 23015654